CLINICAL TRIAL: NCT07258563
Title: Taste Steering in Patients With Cancer Who Are Treated With Chemotherapy: a Multicentre Randomized Intervention Trial
Brief Title: The TASTY-steering Study
Acronym: TASTY-steering
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20862
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Triple Negative Breast Cancer or Metastatic Testicular Cancer, or Stage II-IV Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Testicular Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taste steering (Experimental): To examine the effect of at-home taste steering versus standard care on food enjoyment, the obtained results and outcomes will be measured 1) at baseline before chemotherapy is started, 2) at week 0 when taste or smell alterations occur, and 3) after 6 weeks. The taste steering will take place at home.
  Interventions: Behavioral: Taste steering
- No intervention (No Intervention): standard of care

INTERVENTIONS:
Behavioral: Taste steering — To examine the effect of at-home taste steering versus standard care on food enjoyment, the obtained results and outcomes will be measured 1) at baseline before chemotherapy is started, 2) at week 0 when taste or smell alterations occur, and 3) after 6 weeks. The taste steering will take place at home. The control group will receive usual care. Questionnaires will be filled in online at home, while taste and smell tests and saliva collection will be conducted either at home or in the hospital during regular visits. Patients in both study arms are contacted by their dietitian every 3 weeks.
  Arms: Taste steering

SUMMARY:
This is a multicentre non-blinded randomised intervention trial with a parallel cluster design. The multicentre study will be performed at 12 hospitals in the Netherlands. A parallel cluster design per hospital was selected to prevent contact between participants in the same hospital who are randomised into different study arms. Such contact may result in bias as it may allow for patients in the control arm to be informed about elements of taste steering.

To examine the effect of at-home taste steering versus standard care on food enjoyment, the obtained results and outcomes will be measured 1) at baseline before chemotherapy is started, 2) at week 0 when taste or smell alterations occur, and 3) after 6 weeks. The taste steering will take place at home. The control group will receive usual care. Questionnaires will be filled in online at home, while taste and smell tests and saliva collection will be conducted either at home or in the hospital during regular visits. Patients in both study arms are contacted by their dietitian every 3 weeks.

Some hospitals have implemented elements of taste steering. However, these elements are focused on patients who are admitted to the hospital, and therefore only interfere to a limited extent with the present study that is directed at patients managing their taste alterations at home. Experience with the Smaakpupil tool indicates that the algorithm reaches saturation after 3-4 weeks. Therefore, an intervention period of 6 weeks has been selected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years
* Indication to start chemotherapy for:

  * Metastatic triple negative breast cancer
  * Metastatic testicular cancer
  * Stage II-IV diffuse large B cell lymphoma
* Chemotherapy scheduled to start in the next 6 weeks
* Consuming solid foods and drinks is possible
* ≤50% of recommended daily intake in kcal consists of oral nutritional supplements
* Oral mucositis grade ≤2 (Common Terminology Criteria for Adverse Events, version 5.0)
* Ability to comply with all protocol-required actions
* Written informed consent
* For the intervention phase only: subjective change in taste since start of chemotherapy

Exclusion Criteria:

* Pregnancy
* Currently experiencing taste or smell problems
* Previous or current radiotherapy of head and neck region
* Enteral feeding through tube or parenteral feeding
* Participation in another clinical trial aimed at preventing or treating taste and/or smell alterations
* Chronic (>1 month) high dose corticosteroids (>10 mg prednisone/day or equivalent).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Food enjoyment | 6 weeks
  Food enjoyment, measured by the subsection of the Appetite, Hunger and Sensory Perception Questionnaire (AHSP) after 6 weeks of taste steering compared with standard care

SECONDARY OUTCOMES:
Food enjoyment and liking | 6 weeks
  Food enjoyment and food liking: questions on food enjoyment and food liking on 9-point hedonic scale
Quality of life | 6 weeks
  Quality of life: EORTC QLQ-C30
Taste and smell alterations | 6 weeks
  Taste and smell alterations: Chemotherapy-induced Taste Alteration Scale (ciTAS-NL)
Risk of malnutrition | 6 weeks
  Risk of malnutrition: Patient-Generated Subjective Global Assessment (PG-SGA)
Dry mouth feeling | 6 weeks
  Dry mouth feeling: Xerostomia Inventory (XI) and Regional Oral Dryness Inventory (RODI)
Taste and smell function | 6 weeks
  Taste and smell function
Saliva secretion | 6 weeks
  Saliva secretion
Body weight | 6 weeks
  Body weight

CONTACTS AND LOCATIONS:
Overall Officials: J. J. de Haan, MD, PhD, Principal Investigator — University Medical Center Groningen, Dept. of Medical Oncology
Locations (11):
- Netherlands (11):
  - Amsterdam UMC, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Van Weel-Bethesda Ziekenhuis, Dirksland
  - Ziekenhuisvoorzieningen Gelderse Vallei, Ede
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Radboud University Medical Center, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - Ommelander Ziekenhuis Groningen, Scheemda
  - Maxima Medisch Centrum, Veldhoven
  - Isala Klinieken, Zwolle